CLINICAL TRIAL: NCT01308853
Title: An Open, Multi-center Study Evaluating Treatment Procedure, Efficacy and Safety of Macrolane VRF30 for Enhancement of the Shape and Fullness of the Female Breast
Brief Title: Macrolane for Enhancement of the Shape and Fullness of the Female Breast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31GB0607
Record Dates: First submitted 2011-02-22; First posted 2011-03-04 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2019-06

CONDITIONS: Breast Enhancement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macrolane (Other): Open label
  Interventions: Device: Macrolane

INTERVENTIONS:
Device: Macrolane — Device: Macrolane Treatment: Initial injection (incl touch-up) of a maximum of 120 ml/breast.

SUMMARY:
The study evaluates treatment procedure, efficacy and safety of Macrolane for female breast enhancement.

DETAILED DESCRIPTION:
This study evaluates the injection technique and treatment outcome by stepwise inclusion and treatment of Macrolane for female breast enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Female between 25 and 50 years of age with small breasts seeking enhancement of the shape and fullness of the breast

Exclusion Criteria:

* Unreasonable expectations
* Any medical condition that may interfere with the treatment

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Heden, M.D., Principal Investigator — Akademikliniken, Stockholm, Sweden

REFERENCES:
- [Result] Heden P, Olenius M, Tengvar M. Macrolane for breast enhancement: 12-month follow-up. Plast Reconstr Surg. 2011 Feb;127(2):850-860. doi: 10.1097/PRS.0b013e318200ae57. PMID 20966812

RESULTS

PARTICIPANT FLOW:
Groups:
- Macrolane: Open label
  Device: Macrolane. Treatment: Initial injection (including touch-up) of a maximum of 120 ml/breast.
Period: Overall Study
Arm/Group | Macrolane
Started | 24
Completed | 20
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Insertion of permanent implants | 1

BASELINE CHARACTERISTICS:
Arm/Group | Macrolane
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Breasts With Successful Placement of the Implant Posterior to the Mammary Gland at 6 Weeks After Treatment
Description: Inclusion was made in steps in group of 4 subjects. The subjects were followed-up with MRI 1-5 days after the injection to document correct injection technique. Before the next group were treated, the Expert Group evaluated the 6-week follow-up results of the previous group. The injection procedure was, if necessary, changed in accordance with specifically pre-defined parameters.
Time Frame: 6 weeks
Population: All included participants (Intention To Treat)
Measure: Number; unit: Breasts
Units Other Than Participants: Breasts
Arm/Group | Macrolane
Number analyzed (Participants) | 24
Number analyzed (Breasts) | 48
Breasts | 48

2. Secondary Outcome: Percentage of Breasts With Improvement as Assessed by the Investigator
Description: Esthetic improvement was evaluated using the Global Esthetic Improvement Scale (GEIS).
  The scale has five grades ranging from worse to very much improved. Subjects defined as "at least improved" are assessed as improved, much improved or very much improved.
Time Frame: 6 weeks
Population: Intention to treat. Data from 1 participant not available.
Measure: Number; unit: percentage of breasts
Units Other Than Participants: breasts
Arm/Group | Macrolane
Number analyzed (Participants) | 23
Number analyzed (breasts) | 46
percentage of breasts | 100

ADVERSE EVENTS:
Time Frame: From day 0 up until 24 months after injection
Description: Systematic assessments:
  Subject diary for collection of expected adverse events. Collection of related and unrelated adverse events at each clinical visit following injection when subjects were asked "Since your last clinical visit have you had any health problems?" Mammography performed. Breast examinations Laboratory assessments
Arm/Group | Macrolane
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 18/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macrolane (N=24)
Breast Tenderness (Reproductive system and breast disorders) | 6 (10)
Capsular contracture associated with breast implant (General disorders) | 7 (22)
Injection site pain (General disorders) | 2 (3)
Implant site nodule (General disorders) | 8 (10)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Breast discomfort (Reproductive system and breast disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual publications shall not be made prior to the first, multi-center publication of the results of the multicenter study. The Investigator shall have the right to publish the results of his work. Any publication or presentation by Institution and/or Principal Investigator shall be submitted to Q Med for review and comment no less than 60 days before submission to allow Q Med to determine whether any patentable invention or Confidential Information would be disclosed.